CLINICAL TRIAL: NCT01655095
Title: Improving Bowel Preparation for the Colon Capsule: Picosalax and Prucalopride vs. PEG and Prucalopride
Brief Title: Improving Bowel Preparation for the Colon Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Hotel Dieu Hospital (Gastrointestinal Diseases Research Unit) (Unknown)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DMED-1478-12
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-09

CONDITIONS: Quality of Bowel Preparation for the Colon Capsule; Colon Capsule Completion Rates; Colon Capsule Polyp Detection
Keywords: Colon capsule; Picosalax; PEG; Prucalopride
MeSH Terms: interventions — prucalopride; Bisacodyl; Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG and Prucalopride (Experimental)
  Interventions: Drug: PEG; Drug: Prucalopride; Procedure: Colon capsule; Procedure: Colonoscopy
- Picosalax and Prucalopride (Experimental)
  Interventions: Drug: Prucalopride; Drug: Picosalax; Drug: Bisacodyl; Procedure: Colon capsule; Procedure: Colonoscopy

INTERVENTIONS:
Drug: PEG — PEG 2L at 1800hrs the night before the test and 2L at 0500hrs the morning of the test.
  Arms: PEG and Prucalopride
Drug: Prucalopride — Prucalopride 2mg will be administered at 0800hrs on the day of the test, at the same time the colon capsule is administered. Two hours later the position of the colon capsule will be assess with a Realtime Viewer. If the capsule has not reached the cecum a second dose of Prucalopride 2mg will be administered at that time.
Drug: Picosalax — One sachet at 1800hrs the night before the test One sachet at 0500hrs the day of the test
  Arms: Picosalax and Prucalopride
Drug: Bisacodyl — Bisacodyl 10mg in the evening three nights before the procedure and 10mg again two nights before the procedure.
  Arms: Picosalax and Prucalopride
Procedure: Colon capsule — The colon capsule will be ingested at 0800hrs the day of the test. Seven hours will be allowed for the capsule to clear the bowel. The images will be reviewed by two endoscopists with experience reading video capsule endoscopy.
Procedure: Colonoscopy — At 1500hrs on the day of the test all individuals will return to the endoscopy unit for a colonoscopy.

SUMMARY:
Colon capsule endoscopy is a technology that has been developed as a noninvasive method of examining the large bowel. The biggest limitation to its use has been finding a bowel preparation that will both clean the colon adequately for good visualization of the mucosa and also help propel the capsule through the colon. Most studies have been conducted in Europe using bowel preparation medications that are not approved for use in North America.

The purpose of this study is to compare a combination of polyethylene glycol (PEG) and prucalopride to Picosalax and prucalopride to determine which regime will give a better colon cleanse for the colon capsule. Both PEG and Picosalax are bowel preparations that are used routinely for colonoscopy in Canada. Prucalopride is a new medication recently approved for use in Canada which improves intestinal motility and should help with colon capsule transit.

Patients who are being referred for colonoscopy will be enrolled in the study and randomized to one of the bowel preparation regimes. They will undergo a split-dose bowel preparation with either PEG or Picosalax, which is routine for colonoscopy. As part of the standard bowel preparation, patients randomized to the Picosalax group will take dulcolax three nights before the test and then again two nights before the test. The evening before the test patients will take either PEG 2L or one sachet of Picosalax. The following morning they will take another dose of either PEG (2 Liter container) or one sachet of Picosalax. They will then ingest the colon capsule and a dose of Prucalopride that morning. After 7 hours they will return to the endoscopy unit where they will undergo a colonoscopy, which is the standard of care for examination of the colon.

The images from the colon capsule will be reviewed and the quality of bowel preparation will be graded using a previously validated scale. It is hypothesized that the Picosalax and prucalopride regime will give a better cleanse for the colon than PEG and prucalopride as there will be less turbid fluid in the colon and allow for a better view of the mucosa. Polyp detection and abnormalities of the mucosa detected with the colon capsule will also be compared to polyps and abnormalities detected at the time of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 75
* Patients being referred for colonoscopy

Exclusion Criteria:

* Symptoms of dysphagia
* Bowel obstruction or ileus
* Known stricture or fistula
* Inflammatory bowel disease
* Previous small or large bowel surgery
* Severe gastroparesis or motility disorder
* Renal impairment (GFR<55 within 3 months of study)
* Congestive heart failure (NYHA III or IV)
* Ischemic heart disease
* Cirrhosis or severe hepatic dysfunction (ascites or lab result INR>2)
* History of serious arrhythmia
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the Quality of the Bowel Preparation using a previously defined scale. | Assessed at the time of review of the colon capsule images (from ingestion of capsule until the capsule is passed or the battery runs out--max 10 hrs) and at the time of colonoscopy on the same day (using a previously defined scale as described)
  Cleansing Scale:
  * Poor: Mucosa obscured by opaque debris or turbid fluid
  * Fair: Portion of the mucosa obscured by turbid fluid and/or debris preventing visualization of polyps >5mm in size
  * Good: Fluid was clear and small pieces of debris not obscuring polyps >5mm
  * Excellent: Fluid was clear and either free of debris or only small pieces
  Bubble effect scale:
  * Significant: Bubbles interfere with the examination, >10% surface area obscured by bubbles.
  * Insignificant: No bubbles or bubbles that do not interfere with the examination, <10% of surface area obscured by bubbles.
Number of individuals who have a complete colon capsule study (ie. pass the colon capsule prior to colonoscopy) | Assessed during the time of colon capsule image review

SECONDARY OUTCOMES:
Assessment of patient tolerance of the bowel preparations. | Assessed at the time of colon capsule ingestion (will cover time period from beginning of bowel preparation, as previously described, to ingestion of the colon capsule)
  Survey questionnaire to be completed by participants at the time of the colon capsule endoscopy assessing the tolerability of the preparation and side effects.
Gastric emptying and small and large bowel transit time | Assessed at the time the colon capsule images are reviewed (will be monitored from time of capsule ingestion until capsule is expelled or battery runs out--max 10 hours)
  Determining the amount of time was required for the capsule to transit through the stomach, small bowel and large bowel for the two different preparations based on the images collected during the study.
Comparison of accurate identification of mucosal changes (ie. inflammation) and polyp detection with colonoscopy. | Determined at the time of review of the colon capsule images (assessed from time of capsule ingestion until capsule is expelled or battery runs out--max. 10 hours) and assessed during the colonoscopy the same day.
  Abnormalities identified at the time the colon capsule images are reviewed will be compared to the abnormalities identified during the time of colonoscopy documented in the colonoscopy report.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, Principal Investigator — Queens University; Darlene Brady, Study Director — Queens University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada